CLINICAL TRIAL: NCT04321824
Title: Effectiveness of an Innovative Program in Primary Care for Vulnerable and Precarious Population With Access Barriers to Healthcare System: PASS de Ville
Acronym: EFFIPASS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-23
Record Dates: First submitted 2019-07-10; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-07

CONDITIONS: Vulnerable and Precarious Poupulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the innovative programm (PASS de ville): specific care for precarious people
- the standard of care

SUMMARY:
Since the end of 2018, the Care and Orientation Center (CASO)of Marseille corridnated by Medecins du Monde has been investigated an innovative program aimed at direct referrals to primary care for vulnerable and precarious population with access barriers to healthcare system (no being coveraged at time of the study).

Patients consulting at the CASO MDM in Marseille are accompanied and were received, free of charge, by primary care professionals (general practitioners, specialists, pharmacy, analysis laboratory, etc).

This is an observational, comparative study, with two arms: the CASO MDM in Marseille for the intervention site and the CASO MDM in Bordeaux for the control site (where the innovative program does not exist).

A total of 610 patients will be included (305 in the innovative group / 305 in the control group).

The main objective is to evaluate the effectiveness of the innovative programm (PASS de ville) compared to the standard of care by assessing the rate of emergency departement visits at one year in each group.

Duration of inclusion: 12 months; Duration of follow-up: 18 months; Total duration of the study: 36 months.

Both quantitative and qualitative analyses will be conducted to address overall outcomes.

Univariate and multivariate analyzes will be performed on the primary outcome as well as the secondary outcomes in order to highlight significant differences between the two groups and to identify predictive factors for improved effectiveness. The analysis will be conducted in accordance with Good Epidemiological Practices, and the final report will be written according to the CONSORT (Consolidated Standards of Reporting Trials) recommendations. An intention to treat analysis will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* without health coverage
* having medical needs
* not presenting a vital emergency
* not requiring hospital technical platform
* having declared to want to stay in the area at least 18 months afetr inclusion in the study
* having signed the notice of non opposition to the study

Exclusion Criteria:

* less than 18 years old
* having effective health coverage
* in a life-saving emergency
* needing access to the hospital technical platform
* presenting cognitive impairment that limits comprehension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: vulnerable and precarious population with access barriers to healthcare system ( no being coveraged at time of the study)
Sampling Method: Non-Probability Sample
Enrollment: 488 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
rate of emergency departement visits | 12 months

SECONDARY OUTCOMES:
Mean change from baseline in Quality of life scores on the WHOQOL | 18 months
  WHOQOL scale

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — AP-HM
Locations (1):
- Service Epidémiologie et Economie de la Santé - AP-HM, Marseille, France